CLINICAL TRIAL: NCT05110105
Title: Exploring the Effect of Interactive Board Game Health Education on Improving Stroke Knowledge and Health Literacy in Community-Dwelling Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Li-Fong Lin, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202108063
Record Dates: First submitted 2021-10-13; First posted 2021-11-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive interactive board game health education.
  Interventions: Behavioral: Interactive board game health education
- Control (Active Comparator): Participants will receive conventional health education.
  Interventions: Behavioral: Conventional health education

INTERVENTIONS:
Behavioral: Interactive board game health education — The interactive board game includes risk factors, symptoms, and acute management of stroke. It's a card game combined with (1) addition and subtraction game (risk factors). (2) gestures game (symptoms) (3) matching game (acute management), but in traditional Chinese. The game was implemented in a group (2~6 individuals) for 40 minutes.
  Arms: Intervention
Behavioral: Conventional health education — The health education flier was made refer to medical institutions, e.g., hospitals or clinics, the stroke prevention video was collected from the internet. Participants were assigned to read the health education flier for 20 minutes. Then watch the stroke prevention video for 20 minutes.
  Arms: Control

SUMMARY:
The purpose of this study is to explore the effectiveness between interactive board game health education and conventional health education in improving community-dwelling adults' stroke knowledge and self-reported stroke health literacy, including risk factors, symptoms, acute management of stroke, and 6 aspects of self-reported stroke health literacy. The intervention group will receive an interactive board game in a group (2~6 individuals), while the control group was assigned to read the health education flier and watching the stroke prevention video. The follow-up period was set to be four weeks after the intervention, both control group, and intervention group.

DETAILED DESCRIPTION:
Stroke is a major health problem and a known cause of death and disability. Approximately 13 million people suffered from stroke worldwide annually and it ranks fourth among the top 10 causes of death in Taiwan. In a recent survey of Taiwanese citizens on the World Stroke Day event (New Taipei City) in 2012, the public's stroke literacy was low, only 5.71% of them can reach "good stroke literacy". Generally, stroke education was mostly implemented in a one-way lecture way. Therefore, instead of one-way style health education, the investigators assume that interactive board games can increase stroke knowledge, stroke literacy, and self-reported stroke health literacy of community-dwelling seniors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years old or above.
* Cases with sanity and ability to communicate in Chinese or Taiwanese.
* No oral difficulties in daily life, able to fully express research-relevant narratives and readings.

Exclusion Criteria:

* Patients with a history of stroke diagnosed by a physician.
* Non-Republic of China (Taiwan) nationality.
* Worked as a medical staff in the past, in the fields of medical care or health educator.
* Those who cannot complete the assessment according to the guidance of the assessor.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Stroke Knowledge and Literacy right after the intervention. | Right after the intervention
  Participants' stroke knowledge and literacy were assessed by a questionnaire. Good stroke literacy was determined according to fulfillment of the following criteria: (1) the brain was recognized as the main damaged organ; (2) at least five risk factors of stroke were identified; (3) more than five stroke symptoms were identified; and (4) in case of a stroke, the identified appropriate response was to call 119 immediately. For risk factors and symptoms, according to each correct answer given, a score of either 0 or 1 is given, 1 being the right answer given. A higher score would indicate a better knowledge of the risk factors and symptoms of stroke.
Change from Baseline Stroke Knowledge and Literacy at 4 weeks. | 4 weeks after the intervention
  Participants' stroke knowledge and literacy were assessed by a questionnaire. Good stroke literacy was determined according to fulfillment of the following criteria: (1) the brain was recognized as the main damaged organ; (2) at least five risk factors of stroke were identified; (3) more than five stroke symptoms were identified; and (4) in case of a stroke, the identified appropriate response was to call 119 immediately. For risk factors and symptoms, according to each correct answer given, a score of either 0 or 1 is given, 1 being the right answer given. A higher score would indicate a better knowledge of the risk factors and symptoms of stroke.

SECONDARY OUTCOMES:
Change from Baseline Self-reported Stroke Health Literacy right after the intervention. | Right after the intervention
  Participants' self-reported stroke health literacy was assessed by a questionnaire. The questionnaire contains 6 aspects of stroke health literacy, including the ability to (1) obtain stroke health information; (2) understand written stroke health information; (3) understand oral stroke health information, (4) communicate and being interactive with stroke health information; (5) evaluate and judge stroke health information; (6) apply stroke health information for medical decision-making. A higher score would indicate a better self-reported stroke health literacy.
Change from Baseline Self-reported Stroke Health Literacy at 4 weeks. | 4 weeks after the intervention
  Participants' self-reported stroke health literacy was assessed by a questionnaire. The questionnaire contains 6 aspects of stroke health literacy, including the ability to (1) obtain stroke health information; (2) understand written stroke health information; (3) understand oral stroke health information, (4) communicate and being interactive with stroke health information; (5) evaluate and judge stroke health information; (6) apply stroke health information for medical decision-making. A higher score would indicate a better self-reported stroke health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Da-an Elderly Service and Day Care Center, Taipei, Taiwan